CLINICAL TRIAL: NCT01137734
Title: Valtech Cardinal Adjustable Semi-Rigid Annuloplasty Ring System For Treatment of Mitral Valve Regurgitation in Open Surgical Repair
Brief Title: CARDINAL Adjustable Annuloplasty Ring System For Treatment of Mitral Regurgitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VC1-1
Record Dates: First submitted 2010-05-24; First posted 2010-06-04 (Estimated); Last update posted 2021-11-05 (Actual); Status verified 2021-10

CONDITIONS: Mitral Valve Insufficiency
Keywords: Heart Diseases; Heart Valve Diseases; Cardiovascular Diseases
MeSH Terms: conditions — Mitral Valve Insufficiency; Heart Diseases; Heart Valve Diseases; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Valtech Cardinal Mitral Annuloplasty Ring (Experimental): All subjects enrolled in the study are implanted with the Valtech Cardinal Mitral Annuloplasty ring.
  Interventions: Device: Adjustable Annuloplasty Ring with option to adjust off pump.; Device: Device: Adjustable Annuloplasty Ring (with option to adjust off-pump)

INTERVENTIONS:
Device: Adjustable Annuloplasty Ring with option to adjust off pump. — Annuloplasty device repair of mitral valve regurgitation with option to adjust device post implant off pump, to optimize correction of mitral regurgitation. Unlike conventional annuloplasty repair, the Cardinal system offers the clinician the opportunity to make adjustments after weaning from cardiopulmonary bypass. Adjustability is expected to reduce the number of patients leaving the operating room with residual regurgitation after mitral valve repair.
  Other Names: Valtech Cardinal Adjustable ring
Device: Device: Adjustable Annuloplasty Ring (with option to adjust off-pump) — Evaluate the performance and safety of the investigational adjustable annuloplasty ring device for the treatment of mitral regurgitation, with option to adjust on and off-pump.

SUMMARY:
Annuloplasty device for repair of mitral valve regurgitation with option to adjust device post implant off pump, to optimize correction of mitral regurgitation. Unlike conventional annuloplasty ring, the Cardinal system offers the clinician the opportunity to make adjustments after weaning from cardiopulmonary bypass. Adjustability is expected to reduce the number of patients leaving the operating room with residual regurgitation after mitral valve repair.

ELIGIBILITY:
Inclusion Criteria:

* Patient is a candidate for mitral valve repair.
* Patient able and willing to return to the implant center for follow-up visits.
* Able and willing to give informed consent and follow protocol procedures.

Exclusion Criteria:

* Severe organic lesions with retraction of chordate tendineae, severly fibrotic and immobile leaflets, severely deformed subvalvular apparatus.
* Evolving endocarditis or active endocarditis in the last 3 months.
* Heavily calcified annulus or leaflets.
* Congenital malformation with limited valvular tissue
* Patient requires mitral valve replacement.
* Previously implanted prosthetic mitral valve or annuloplasty ring/band.
* Patient requires aortic or pulmonic valve replacement or repair.
* Patient is pregnant (urine HCG test result positive) or lactating.
* Patient has a major cardiac or non-cardiac disease, which in the investigator's experience produces an unacceptable surgical risk.
* Life expectancy of less than twelve months.
* Patient is participating in concomitant research studies of investigational products

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-03; Primary Completion 2012-02 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Percentage of Subjects with Valtech Cardinal Mitral Heart Valve Device Technical Success | Day of surgery
  Technical success of the implantation of the Cardinal Ring defined as the ability to size the annulus, place the sutures on the ring, lower the ring onto the valve, adjust the ring to the required size and disconnect the adjustment tool.
Percentage of Subjects with Successful Off Pump Adjustment of their Valtech Cardinal Mitral Annuloplasty Ring | Day of surgery
  The technical feasibility of "off cardiac bypass pump" adjustment during surgery, when required of the Valtech Cardinal Mitral Heart Valve Annuloplasty Ring.
Subject's Mitral Valve Regurgitation (MR) Post-procedure as Compared to Baseline | At the end of the procedure on the day of surgery compared to baseline.
  The percentage of subjects that had a reduction of their pre-operative mitral regurgitation grade as compared to the mitral regurgitation grade at the end of the procedure with the Valtech Cardinal Mitral Heart Valve Annuloplasty Ring.
Subject's Mitral Valve Regurgitation (MR) at Discharge as Compared to Baseline | Day of discharge compared to baseline.
  The percentage of subjects that had a reduction of their pre-operative mitral regurgitation grade as compared to the mitral regurgitation grade at hospital discharge with the Valtech Cardinal Mitral Heart Valve Annuloplasty Ring.
Subject's Mitral Valve Regurgitation (MR) at 30 Days as Compared to Baseline | 30 days compared to baseline.
  The percentage of subjects that had a reduction of their pre-operative mitral regurgitation grade as compared to the mitral regurgitation grade at 30 days with the Valtech Cardinal Mitral Heart Valve Annuloplasty Ring.

SECONDARY OUTCOMES:
Subject's Device Related Adverse Event Rate | 6 months
  The percentage of subjects that had a device related adverse event with the Valtech Cardinal Mitral Heart Valve Annuloplasty Ring.

CONTACTS AND LOCATIONS:
Overall Officials: Hugo Vanermen, Prof, MD, Principal Investigator — Hospital Onze-Lieve-Vrouw-Ziekenhuis, Aalst , Belgium; Fredrich Mohr, Prof,MD, Principal Investigator — University Leipzig, Germany; Volkmar Falk, Prof, MD, Principal Investigator — University Zurich, Switzerland
Locations (2):
- Hugo Vanermen, Aalst, Belgium
- Hospital San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be available to other researchers.

REFERENCES:
- [Background] Si MS, Conte JV, Romano JC, Romano MA, Andersen ND, Gerdisch MW, Kupferschmid JP, Fiore AC, Bakhos M, Bonilla JJ, Burke JR, Rankin JS, Wei LM, Badhwar V, Turek JW. Unicuspid Aortic Valve Repair Using Geometric Ring Annuloplasty. Ann Thorac Surg. 2021 Apr;111(4):1359-1366. doi: 10.1016/j.athoracsur.2020.04.147. Epub 2020 Jun 30. PMID 32619617
- [Background] Czesla M, Gotte J, Voth V, Doll N. Single-Center Experience With Adjustable Annuloplasty Ring in Degenerative Mitral Regurgitation. Innovations (Phila). 2015 Jul-Aug;10(4):248-51; discussion 251. doi: 10.1097/IMI.0000000000000186. PMID 26371453
- [Background] Kolsut P, Juraszek A, Brzozowski P, Dabrowski M, Witkowski A, Rozanski J, Kusmierczyk M. Case report on successful 'bail out' aortic homograft implantation in a 81-year old woman with aortic ring rupture after double TAVI procedure. J Cardiothorac Surg. 2015 Mar 4;10:28. doi: 10.1186/s13019-015-0233-x. PMID 25887519
- [Background] Maisano F, Falk V, Borger MA, Vanermen H, Alfieri O, Seeburger J, Jacobs S, Mack M, Mohr FW. Improving mitral valve coaptation with adjustable rings: outcomes from a European multicentre feasibility study with a new-generation adjustable annuloplasty ring system. Eur J Cardiothorac Surg. 2013 Nov;44(5):913-8. doi: 10.1093/ejcts/ezt128. Epub 2013 Mar 25. PMID 23530026